CLINICAL TRIAL: NCT00217477
Title: An Open Label, Dose Escalation Study of Paricalcitol (Zemplar™) [19-NOR-1 ALPHA, 25-(OH) D] in Combination With Gemcitabine [2', 2' -Difluorodeoxycytidine] in Patients With Advanced Malignancies
Brief Title: Paricalcitol and Gemcitabine in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441212
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paricalcitol IV in combination with Gemcitabine IV (Experimental): Patients receive gemcitabine hydrochloride IV over 80 minutes on days 1, 8, and 15 and paricalcitol IV over 15 minutes on days 7 and 14 in course 1. Beginning in course 2, patients receive paricalcitol IV over 15 minutes on days 1, 8, and 15 and gemcitabine hydrochloride IV over 80 minutes on days 2, 9, and 16. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: paricalcitol

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
Drug: paricalcitol — Given IV

SUMMARY:
RATIONALE: Paricalcitol may cause cancer cells to look more like normal cells, and to grow and spread more slowly. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving paricalcitol together with gemcitabine may be an effective treatment for cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of paricalcitol when given together with gemcitabine in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of paricalcitol when given with gemcitabine in patients with advanced malignancy.

Secondary

* Determine safety and toxicity of this regimen in these patients.
* Determine the pharmacokinetics of these regimens in these patients.
* Determine the clinical outcome (overall survival and best overall response) of patients treated with this regimen.

OUTLINE: This is a dose-escalation, open-label study.

Patients receive gemcitabine IV over 80 minutes on days 1, 8, and 15 and paricalcitol IV over 15 minutes on days 7 and 14 in course 1. Beginning in course 2, patients receive paricalcitol IV over 15 minutes on days 1, 8, and 15 and gemcitabine IV over 80 minutes on days 2, 9, and 16. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paricalcitol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients are treated at the MTD.

After completion of study treatment, patients are followed for survival.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced malignancy

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist or are no longer effective
* No known brain metastases

  * Patients with previously treated brain metastases are eligible provided they have recovered from prior treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 3.0 times upper limit of normal

Renal

* Creatinine ≤ 2.0 mg/dL
* Corrected calcium ≤ 10.5 mg/dL
* Prior single confirmed urolithiasis allowed provided patient is free of stone formation for ≥ 5 years
* No calculi in the urinary tract on kidney ultrasound biopsy or other imaging studies

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* Curative therapy for a condition associated with the risk of renal stones (e.g., hyperparathyroidism, bladder dysfunction, or obstructive uropathy) allowed provided patients have been free of stone formation for ≥ 5 years
* No concurrent digoxin
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-08; Primary Completion 2013-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of i. v. pancalcitol given weekly, in combination with fixed dose rate infusion of i. v.gemcitabine given weekly in patients with advanced malignancies. | 4 weeks

SECONDARY OUTCOMES:
To assess toxicity. | 8 week intervals
To determine the effects of paricalcitol on the pharmacokinetics of gemcitabine. | Days 1 & 8, cycle 1
To determine the effects of pariclcitol on cytidine deaminase in PBM | Days 1 & 8, cycle 1
To determine the effects of paricalcitol on dFdCTP in PBM | Days 1 & 8, cycle 1
To determine the pharmacokinetics of paricalcitol when given with gemcitabine | Day 7, cycle 1
To describe clinical outcome for response and survival | 8 week intervals

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States